CLINICAL TRIAL: NCT02274662
Title: Expanded Access Protocol Thymus Transplantation for Immunodeficiency, Hematologic Malignancies, and Autoimmune Disease Related to Poor Thymic Function
Brief Title: Expanded Access Protocol Thymus Transplantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sumitomo Pharma Switzerland GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00051692
Record Dates: First submitted 2014-10-22; First posted 2014-10-24 (Estimated); Results first posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2024-12

CONDITIONS: Poor Thymic Function; Immunodeficiency; Athymia; Immunoreconstitution; Thymus Transplantation; Low T Cell Numbers
Keywords: Cultured Thymus Tissue Implantation
MeSH Terms: conditions — Immunologic Deficiency Syndromes; Thymic aplasia | interventions — Blood Specimen Collection; Phlebotomy; Antilymphocyte Serum; Cyclosporine; Tacrolimus; Cyclosporins

ARMS (1):
- Cultured thymus tissue implantation (CTTI) (Experimental): Cultured thymus tissue for the treatment of immunodeficiency and autoimmune disorders
  Interventions: Biological: Cultured Thymus Tissue; Procedure: Blood Draw; Drug: Rabbit Anti-Thymocyte Globulin and Cyclosporine or Tacrolimus

INTERVENTIONS:
Biological: Cultured Thymus Tissue — Subjects receive cultured thymus tissue which is implanted into the quadriceps muscle. Subjects may receive pre and/or post-implantation immunosuppression.
  Potential subjects are screened for eligibility. The thymus tissue (from an unrelated donor), the donor, and the donor's mother are screened for safety. Cultured thymus tissue is implanted into the subject's quadriceps muscle under general anesthesia in the operating room. Two to three months post-implantation, if medically stable, subjects may undergo an allograft biopsy. Subjects undergo laboratory testing for approximately one year post-implantation. At year 2 post-implantation, subjects are contacted for data collection.
Procedure: Blood Draw
  Other Names: Venipuncture
Drug: Rabbit Anti-Thymocyte Globulin and Cyclosporine or Tacrolimus — RATGAM and Cyclosporine or Tacrolimus may be given, depending on the patient. The doses, timing, and trough levels will vary depending on the patient's clinical condition.
  Other Names: RATGAM and Csa or FK506

SUMMARY:
The primary purpose is to provide access for patients who have immunodeficiency or severe autoimmune disease related to poor thymic function to cultured thymus tissue for implantation. With no thymus function, bone marrow stem cells do not develop into educated T cells, which fight infection.

Eligible participants receive cultured thymus tissue for implantation and may undergo biopsy. Immune suppression may be given depending on the immune status and clinical condition of the participant. Immune function testing is continued for one year post-implantation.

DETAILED DESCRIPTION:
The patients enrolled have a high likelihood of death if they do not receive culture thymus tissue because of lack of thymus function. As there are many types of patients who may be enrolled, study results will not have statistical significance.

The study objective is to make cultured thymus tissue available for implantation on an expanded access basis. Data will be collected on survival, naïve T cell development, T cell chimerism, and implant related toxicities, as well as any unexpected study-related serious adverse events.

Eligible subjects receive cultured thymus tissue and may undergo allograft biopsy. Immune suppression may be given depending on the subject's immune status and clinical condition.

Protocol specified studies continue until approximately one year post-implantation. Study participation lasts approximately two years.

ELIGIBILITY:
Cultured Thymus Tissue Inclusion Criteria for Implantation:

* an immunodeficiency or severe autoimmunity for which development of naïve T cells would be expected to lead to lead to clinical improvement.
* written consent (or consent of parent/legal guardian as applicable), review of medical testing, laboratory studies, and physical examinations are used to determine whether the patient is clinically stable and will potentially benefit from receiving cultured thymus tissue. Each participant is reviewed with the Data Safety and Monitoring Board (DSMB).

Cultured Thymus Tissue Exclusion Criteria for Implantation:

* Unrepaired cyanotic congenital heart disease
* Uncontrolled infections. "Uncontrolled" is defined as requiring a ventilator, dialysis, or vasopressor support or anticipated as requiring such support within 6 months.
* Pregnancy

  * For females of child-bearing potential, a serum pregnancy test is done after consent, at the same time another blood draw is done if possible.
  * Females of child-bearing potential must agree to contraceptive measures as indicated in the consent form.
  * A second serum pregnancy test is done within 48 hours prior to administration of study interventions involving FDA pregnancy class D drugs, chemotherapy drugs, or other drugs or interventions known to pose risks to a potential fetus.
* HIV Positive
* History of malignancy
* CMV Infection

  * For subjects receiving immunosuppression as part of the implantation protocol, CMV infection as documented by >500 copies/ml in blood by PCR on two consecutive assays is an exclusion.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2023-08 (Actual); Study Completion 2023-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John W. Sleasman, M.D., Principal Investigator — Duke University Medical Center, Pediatrics, Allergy & Immunology

REFERENCES:
- [Background] Markert ML, Devlin BH, Alexieff MJ, Li J, McCarthy EA, Gupton SE, Chinn IK, Hale LP, Kepler TB, He M, Sarzotti M, Skinner MA, Rice HE, Hoehner JC. Review of 54 patients with complete DiGeorge anomaly enrolled in protocols for thymus transplantation: outcome of 44 consecutive transplants. Blood. 2007 May 15;109(10):4539-47. doi: 10.1182/blood-2006-10-048652. Epub 2007 Feb 6. PMID 17284531
- [Background] Markert ML, Devlin BH, McCarthy EA. Thymus transplantation. Clin Immunol. 2010 May;135(2):236-46. doi: 10.1016/j.clim.2010.02.007. Epub 2010 Mar 16. PMID 20236866
- [Background] Markert ML, Alexieff MJ, Li J, Sarzotti M, Ozaki DA, Devlin BH, Sedlak DA, Sempowski GD, Hale LP, Rice HE, Mahaffey SM, Skinner MA. Postnatal thymus transplantation with immunosuppression as treatment for DiGeorge syndrome. Blood. 2004 Oct 15;104(8):2574-81. doi: 10.1182/blood-2003-08-2984. Epub 2004 Apr 20. PMID 15100156
- [Background] Selim MA, Markert ML, Burchette JL, Herman CM, Turner JW. The cutaneous manifestations of atypical complete DiGeorge syndrome: a histopathologic and immunohistochemical study. J Cutan Pathol. 2008 Apr;35(4):380-5. doi: 10.1111/j.1600-0560.2007.00816.x. PMID 18333898
- [Background] Chinn IK, Devlin BH, Li YJ, Markert ML. Long-term tolerance to allogeneic thymus transplants in complete DiGeorge anomaly. Clin Immunol. 2008 Mar;126(3):277-81. doi: 10.1016/j.clim.2007.11.009. Epub 2007 Dec 26. PMID 18155964
- [Background] Markert ML, Li J, Devlin BH, Hoehner JC, Rice HE, Skinner MA, Li YJ, Hale LP. Use of allograft biopsies to assess thymopoiesis after thymus transplantation. J Immunol. 2008 May 1;180(9):6354-64. doi: 10.4049/jimmunol.180.9.6354. PMID 18424759
- [Background] Hudson LL, Louise Markert M, Devlin BH, Haynes BF, Sempowski GD. Human T cell reconstitution in DiGeorge syndrome and HIV-1 infection. Semin Immunol. 2007 Oct;19(5):297-309. doi: 10.1016/j.smim.2007.10.002. Epub 2007 Nov 26. PMID 18035553
- [Background] Markert ML, Devlin BH, Chinn IK, McCarthy EA. Thymus transplantation in complete DiGeorge anomaly. Immunol Res. 2009;44(1-3):61-70. doi: 10.1007/s12026-008-8082-5. PMID 19066739
- [Background] Markert ML, Alexieff MJ, Li J, Sarzotti M, Ozaki DA, Devlin BH, Sempowski GD, Rhein ME, Szabolcs P, Hale LP, Buckley RH, Coyne KE, Rice HE, Mahaffey SM, Skinner MA. Complete DiGeorge syndrome: development of rash, lymphadenopathy, and oligoclonal T cells in 5 cases. J Allergy Clin Immunol. 2004 Apr;113(4):734-41. doi: 10.1016/j.jaci.2004.01.766. PMID 15100681
- [Background] Markert ML, Devlin BH, McCarthy EA, Chinn IK, Hale LP. Thymus Transplantation in Thymus Gland Pathology: Clinical, Diagnostic, and Therapeutic Features. Eds Lavinin C, Moran CA, Morandi U, Schoenhuber R. Springer-Verlag Italia, Milan, 2008, pp 255-267.
- [Background] Markert ML and Devlin BH. Thymic reconstitution (in Rich RR, Shearer WT, Fleischer T, Schroeder HW, Weyand CM, Frew A, eds., Clinical Immunology 3rd edn., Elsevier, Edinburgh) p 1253-1262, 2008.
- [Background] Markert ML, Sarzotti M, Ozaki DA, Sempowski GD, Rhein ME, Hale LP, Le Deist F, Alexieff MJ, Li J, Hauser ER, Haynes BF, Rice HE, Skinner MA, Mahaffey SM, Jaggers J, Stein LD, Mill MR. Thymus transplantation in complete DiGeorge syndrome: immunologic and safety evaluations in 12 patients. Blood. 2003 Aug 1;102(3):1121-30. doi: 10.1182/blood-2002-08-2545. Epub 2003 Apr 17. PMID 12702512
- [Background] Chinn IK, Olson JA, Skinner MA, McCarthy EA, Gupton SE, Chen DF, Bonilla FA, Roberts RL, Kanariou MG, Devlin BH, Markert ML. Mechanisms of tolerance to parental parathyroid tissue when combined with human allogeneic thymus transplantation. J Allergy Clin Immunol. 2010 Oct;126(4):814-820.e8. doi: 10.1016/j.jaci.2010.07.016. Epub 2010 Sep 15. PMID 20832849
- [Background] Markert ML, Marques JG, Neven B, Devlin BH, McCarthy EA, Chinn IK, Albuquerque AS, Silva SL, Pignata C, de Saint Basile G, Victorino RM, Picard C, Debre M, Mahlaoui N, Fischer A, Sousa AE. First use of thymus transplantation therapy for FOXN1 deficiency (nude/SCID): a report of 2 cases. Blood. 2011 Jan 13;117(2):688-96. doi: 10.1182/blood-2010-06-292490. Epub 2010 Oct 26. PMID 20978268
- [Background] Li B, Li J, Devlin BH, Markert ML. Thymic microenvironment reconstitution after postnatal human thymus transplantation. Clin Immunol. 2011 Sep;140(3):244-59. doi: 10.1016/j.clim.2011.04.004. Epub 2011 Apr 16. PMID 21565561
- [Background] Albuquerque AS, Marques JG, Silva SL, Ligeiro D, Devlin BH, Dutrieux J, Cheynier R, Pignata C, Victorino RM, Markert ML, Sousa AE. Human FOXN1-deficiency is associated with alphabeta double-negative and FoxP3+ T-cell expansions that are distinctly modulated upon thymic transplantation. PLoS One. 2012;7(5):e37042. doi: 10.1371/journal.pone.0037042. Epub 2012 May 10. PMID 22590644
- [Background] Markert ML, Devlin BH, Chinn IK, McCarthy EA, Li YJ. Factors affecting success of thymus transplantation for complete DiGeorge anomaly. Am J Transplant. 2008 Aug;8(8):1729-36. doi: 10.1111/j.1600-6143.2008.02301.x. Epub 2008 Jun 28. PMID 18557726
- [Background] Heimall J, Keller M, Saltzman R, Bunin N, McDonald-McGinn D, Zakai E, de Villartay JP, Moshous D, Ariue B, McCarthy EA, Devlin BH, Parikh S, Buckley RH, Markert ML. Diagnosis of 22q11.2 deletion syndrome and artemis deficiency in two children with T-B-NK+ immunodeficiency. J Clin Immunol. 2012 Oct;32(5):1141-4. doi: 10.1007/s10875-012-9741-9. Epub 2012 Aug 3. PMID 22864628
- [Background] Ciupe SM, Devlin BH, Markert ML, Kepler TB. Quantification of total T-cell receptor diversity by flow cytometry and spectratyping. BMC Immunol. 2013 Aug 6;14:35. doi: 10.1186/1471-2172-14-35. PMID 23914737
- [Background] Ciupe SM, Devlin BH, Markert ML, Kepler TB. The dynamics of T-cell receptor repertoire diversity following thymus transplantation for DiGeorge anomaly. PLoS Comput Biol. 2009 Jun;5(6):e1000396. doi: 10.1371/journal.pcbi.1000396. Epub 2009 Jun 12. PMID 19521511
- [Background] Chinn IK, Milner JD, Scheinberg P, Douek DC, Markert ML. Thymus transplantation restores the repertoires of forkhead box protein 3 (FoxP3)+ and FoxP3- T cells in complete DiGeorge anomaly. Clin Exp Immunol. 2013 Jul;173(1):140-9. doi: 10.1111/cei.12088. PMID 23607606
- [Background] Li B, Li J, Hsieh CS, Hale LP, Li YJ, Devlin BH, Markert ML. Characterization of cultured thymus tissue used for transplantation with emphasis on promiscuous expression of thyroid tissue-specific genes. Immunol Res. 2009;44(1-3):71-83. doi: 10.1007/s12026-008-8083-4. PMID 19066738
- [Background] Gupton SE, McCarthy EA, Markert ML. Care of Children with DiGeorge Before and After Cultured Thymus Tissue Implantation. J Clin Immunol. 2021 Jul;41(5):896-905. doi: 10.1007/s10875-021-01044-0. Epub 2021 May 18. PMID 34003433
- [Background] Markert ML, Gupton SE, McCarthy EA. Experience with cultured thymus tissue in 105 children. J Allergy Clin Immunol. 2022 Feb;149(2):747-757. doi: 10.1016/j.jaci.2021.06.028. Epub 2021 Aug 4. PMID 34362576

RESULTS

PARTICIPANT FLOW:
Groups:
- Cultured Thymus Tissue Implantation: Cultured thymus tissue for the treatment of immunodeficiency and autoimmune disorders
Period: Overall Study
Arm/Group | Cultured Thymus Tissue Implantation
Started | 11
Completed | 7
Not Completed | 4
Not completed — Death | 1
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | Cultured Thymus Tissue Implantation
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: days] | 1485.5 (1601.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Survival Rate at End of 1 Year
Time Frame: 1 Year
Population: Efficacy Analysis Set (EAS): EAS set includes all subjects with athymia associated with complete DiGeorge anomaly or FoxN1 deficiency, who had no prior hematopoietic cell transplant (HCT) and were treated with cultured postnatal thymus tissue in study 51692
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cultured Thymus Tissue Implantation
Number analyzed (Participants) | 11
percentage of participants | 90.9 [59 to 100]

2. Primary Outcome: Survival Rate at End of 2 Year
Time Frame: 2 Year
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cultured Thymus Tissue Implantation
Number analyzed (Participants) | 11
percentage of participants | 87.5 [47 to 100]

ADVERSE EVENTS:
Time Frame: 2 years
Description: within 2 Years of Transplantation
Arm/Group | Cultured Thymus Tissue Implantation
All-Cause Mortality (participants affected / at risk) | 1/11
Serious Adverse Events (participants affected / at risk) | 8/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cultured Thymus Tissue Implantation (N=11)
Device related infection (Infections and infestations) | 3 (13)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2)
Bacterial infection (Infections and infestations) | 1 (1)
Bacterial tracheitis (Infections and infestations) | 1 (2)
Clostridium difficile colitis (Infections and infestations) | 1 (2)
Lower respiratory tract infection bacterial (Infections and infestations) | 1 (2)
Respiratory tract infection bacterial (Infections and infestations) | 1 (2)
Tracheitis (Infections and infestations) | 1 (2)
Cellulitis (Infections and infestations) | 1 (1)
Gastroenteritis adenovirus (Infections and infestations) | 1 (1)
Lower respiratory tract infection viral (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Sinusitis fungal (Infections and infestations) | 1 (1)
Subacute endocarditis (Infections and infestations) | 1 (1)
Viraemia (Infections and infestations) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Coombs positive haemolytic anaemia (Blood and lymphatic system disorders) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1)
Histiocytosis haematophagic (Blood and lymphatic system disorders) | 1 (1)
Splenomegaly (Blood and lymphatic system disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Pneumatosis (General disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Graft versus host disease (Immune system disorders) | 1 (1)
Stress fracture (Injury, poisoning and procedural complications) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Thrombosis in device (Product Issues) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cultured Thymus Tissue Implantation (N=11)
Viral upper respiratory tract infection (Infections and infestations) | 2 (4)
Acarodermatitis (Infections and infestations) | 1 (1)
Bacterial infection (Infections and infestations) | 1 (1)
Clostridium bacteraemia (Infections and infestations) | 1 (1)
Ear infection fungal (Infections and infestations) | 1 (1)
Gastroenteritis norovirus (Infections and infestations) | 1 (1)
Oesophageal candidiasis (Infections and infestations) | 1 (1)
Oral viral infection (Infections and infestations) | 1 (1)
Otitis media chronic (Infections and infestations) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1)
Sinusitis bacterial (Infections and infestations) | 1 (1)
Viral rash (Infections and infestations) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (3)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1)
Weight gain poor (Metabolism and nutrition disorders) | 1 (1)
Irritability (Psychiatric disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Left ventricular hypertrophy (Cardiac disorders) | 1 (2)
Hypertension (Vascular disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Gingival hypertrophy (Gastrointestinal disorders) | 1 (1)
Hepatomegaly (Hepatobiliary disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Glycosuria (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Pyrexia (General disorders) | 5 (6)
Oedema peripheral (General disorders) | 1 (1)
Blood creatinine increased (Investigations) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood iron decreased (Investigations) | 1 (1)
Lipase increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Weight decreased (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the event the Study is part of a multi-center study, the first publication of the results of the Study shall be made in conjunction with the results of other participating study sites as a multi-center publication; provided however, if a multi-center publication is not forthcoming within twenty-four (24) months following completion of the Study at all sites, Institution and Investigator shall be free to publish.

DOCUMENTS (2):
  • Study Protocol (2021-11-30): https://cdn.clinicaltrials.gov/large-docs/62/NCT02274662/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-19): https://cdn.clinicaltrials.gov/large-docs/62/NCT02274662/SAP_001.pdf